CLINICAL TRIAL: NCT04615975
Title: Pilot Study: Ketogenic Diet as Protective Factor During SARS-CoV-2 Infection
Brief Title: Ketogenic Diet as Protective Factor During COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Padova (Other)
Collaborators: San Bortolo Hospital - Vicenza (Unknown)
Responsible Party: Principal Investigator, Antonio Paoli, Full Professor, University of Padova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KDSARS0120
Record Dates: First submitted 2020-10-31; First posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Covid19
Keywords: inflammation; cytokines; SARS-CoV-2; Ketogenic diet; ketosis
MeSH Terms: conditions — COVID-19; Inflammation; Ketosis | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Patients will receive 21 days of a very low carbohydrate mediterranean ketogenic diet with phytoextracts and 7 days of a low carbohydrate diet
  Interventions: Dietary Supplement: Ketogenic diet with phytoextracts

INTERVENTIONS:
Dietary Supplement: Ketogenic diet with phytoextracts — Patients were provided with an individualized nutritional ketogenic plan during hospitalization

SUMMARY:
The novel coronavirus disease (COVID-19) is posing a serious challenge to the health-care systems worldwide, with an enormous impact on health conditions and loss of lives. More than 30 millions of recoveries worldwide were registered at the end of October 2020 with more than 1 million of deaths. As the disease continues to spread, strategies aimed to reduce hospitalization time in sub intensive unit care, thus reducing pressure on health system, but also to reduce some of the pathological features of COVID-19 such as inflammation and the "cytokines storm".

The ketogenic diet is a high fat, low carbohydrate, adequate-protein diet that promotes a physiological ketosis (due to an increase of liver ketone bodies production). High fat, low carbohydrate diets have been shown to reduce duration of ventilator support and partial pressure carbon dioxide in patients with acute respiratory failure. Moreover, the physiological increase in plasma levels of ketone bodies exerts important anti-inflammatory and immunomodulating effects, which may reveal as precious tools to reduce potential adverse outcomes of COVID-19 disease.

The hypothesis of this study is that the administration of a ketogenic diet will improve gas exchange, reduce inflammation, and the duration of hospitalization. The plan is to enrol 28 patients with diagnosis of COVID-19 hospitalized but not in ICU with SPO2 higher than 88%.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized Hospital with COVID-19 diagnosis (nasopharyngeal and oropharyngeal swab)
* peripheral oxygen saturation higher tha 88%

Exclusion Criteria:

* intensive unit care
* under forced ventilation
* peripheral oxygen saturation lower than 88%
* parenteral nutrition

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
inflammation panel: interleukine 6 (IL-6) | Daily until patient's hospital discharge, up to 30 days
  change in IL-6 levels. IL-6 is an inflammatory cytokine. Units: in pg/mL
inflammation panel: tumor necrosis factor alfa (TNFα) | Daily untilpatient's hospital discharge, up to 30 days
  change in TNFα levels. TNFα is an inflammatory cytokine Units: pg/mL
inflammation panel: C-reactive Protein (CRP) | Daily until patient's hospital discharge, up to 30 days
  change in CRP levels. CRP is an non specific index of inflammation Units: in mg/dL
inflammation panel: Erythrocyte sedimentation rate (ESR) | Daily untilpatient's hospital discharge, up to 30 days
  change in ESR. ESR is an non specific index of inflammationUnits: mm/h
coagulation panel: D-Dimer | Daily until patient's hospital discharge, up to 30 days
  change in D-Dimer levels. D-Dimer is a fibrin degradation product. Units: 0.5 mcg/ml Fibrinogen Equivalent Units (FEU)
coagulation panel: fibrinogen | Daily until patient's hospital discharge, up to 30 days
  change in fibrinogen levels. Fibrinogen is a protein involved in forming blood clots in the body. Units: mg/dL
coagulation panel: thrombin clotting time (TT) | Daily until patient's hospital discharge, up to 30 days
  change in TT. TT measures the time it takes for a clot to form in the plasma of a blood sample containing anticoagulant, after an excess of thrombin has been added. Units: seconds
coagulation panel: activated partial thromboplastin time (aPTT) | Daily until patient's hospital discharge, up to 30 days
  change inl aPTT. aPTT measures the overall speed at which blood clots by means of two consecutive series of biochemical reactions. Units: in seconds
Dyspnoea Visual Analog Scale Score (VAS) | Daily until patient's hospital discharge, up to 30 days
  Change in VAS. VAS is a horizontal line, 100 mm in length, and anchored by word descriptors at each end. The VAS dyspnea score uses "no shortness of breath at all" and "maximum shortness of breath". The patient marks on the line the point that they feel represents the perception of their current state
Oxygen saturation | Continuosly, daily until patient's hospital discharge, up to 30 days
  change in basal peripheral oxygen saturation percentage (%)
Evaluation of Lungs conditions | Change from baseline, Every three days until patient's hospital discharge, up to 30 days
  Anteroposterior chest radiography (CXR)
The total hospital stay | up to 30 days
  Time from hospital admission to discharge from the hospital.

SECONDARY OUTCOMES:
Mean Corpuscular Hemoglobin (MCH) | Daily until patient's hospital discharge, up to 30 days
  Change in the amount of hemoglobin per red blood cell. Mean cell hemoglobin is the average mass of hemoglobin per red blood cell in a sample of blood. Units: picograms (pg) per cell
Mean corpuscular volume (MCV) | Daily until patient's hospital discharge, up to 30 days
  change in the size of the red blood cells. Mean cell volume is a measure of the average volume of a red blood corpuscle. Units: femtoliters
mean corpuscular hemoglobin concentration (MCHC) | Daily until patient's hospital discharge, up to 30 days
  change in the amount of hemoglobin per unit volume. Mean cell hemoglobin concentration is the average concentration of hemoglobin in a given volume of blood. Unites: g/dl of red blood cells
haemoglobin Hb | Daily until patient's hospital discharge, up to 30 days
  change in total hemoglobin. Hemoglobin is an indirect way to measure red blood cells. Units: g/ dL
Red blood cells count | Daily until patient's hospital discharge, up to 30 days
  Change in the number of red blood cells. Red blood cell count measure anemia. Units: million cells per microliter (cells/mcL)
beta - hydroxybutyrate (BHB) | Daily until patient's hospital discharge, up to 30 days
  Change in ketonemia measured as concentration of blood BHB Units: mmol/L
Alanine transaminase (ALT) | Daily until patient's hospital discharge, up to 30 days
  Change in ALT. ALT is a liver function test. Units: mU/ml
Aspartate transaminase (AST) | Daily until patient's hospital discharge, up to 30 days
  Change in AST. AST ALT is a liver function test. Units : mU/ml
lactate dehydrogenase (LDH) | Daily until patient's hospital discharge, up to 30 days
  Change in LDH. LDH is a marker of tissues damage. Units: Unites/L

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Paoli, MD, Principal Investigator — University of Padova
Locations (1):
- Ospedale San Bortolo, Vicenza, Italy